CLINICAL TRIAL: NCT02607683
Title: A Phase 2b/3, Multicenter, Dose-ranging, Randomized, Double-masked, Placebo-controlled Study of XAF5 Ointment for Reduction of Lower Lid Steatoblepharon
Brief Title: Phase 2b/3 Study of XAF5 Ointment for Steatoblepharon (Undereye Bags)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XOPH5-OINT-3
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Steatoblepharon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- XAF5 (concentration A: 0.1%) (Experimental): Participants will apply XAF5 Ointment (concentration A: 0.1%) to the lower eyelids once daily.
  Interventions: Drug: XAF5 (concentration A: 0.1%)
- XAF5 (concentration B: 0.035%) (Experimental): Participants will apply XAF5 Ointment (concentration B: 0.035%) to the lower eyelids once daily.
  Interventions: Drug: XAF5 (concentration B: 0.035%)
- Placebo (Placebo Comparator): Participants will apply Placebo Ointment to the lower eyelids once daily.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: XAF5 (concentration A: 0.1%)
  Arms: XAF5 (concentration A: 0.1%)
Drug: XAF5 (concentration B: 0.035%)
  Arms: XAF5 (concentration B: 0.035%)
Drug: Matching placebo
  Arms: Placebo

SUMMARY:
This randomized, placebo-controlled, double-masked, Phase 2b/Phase 3 study will assess the efficacy of two different concentrations of XAF5 Ointment for reduction of lower lid steatoblepharon (undereye bags).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe, bilateral lower eyelid steatoblepharon
* Must understand and provide informed consent
* Healthy facial skin

Exclusion Criteria:

* Pregnant or lactating women
* Clinically significant eye disease
* Best corrected visual acuity worse than 20/40 in either eye
* History of eye surgery in past 6 months
* History of lower eyelid surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
LESS score (Clinician-Reported) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie Roth, Ph.D., Study Director — Allergan
Locations (6):
- United States (6):
  - David Wirta, MD, Inc., Newport Beach, California
  - OC Clinical Trials, Santa Ana, California
  - Danbury Eye Physicians, Danbury, Connecticut
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - South Shore Eye Care, Inc., Wantagh, New York
  - Cincinatti Eye Institute, Cincinnati, Ohio